CLINICAL TRIAL: NCT06925971
Title: A Prospective, Multi-center, Open-label, Controlled, Superiority, Randomized, Controlled Registration Trial of the Rapamycin Target Eluting Stent for the Treatment of Symptomatic Cerebral Artery Atherosclerotic Disease（TARGET-DREAM）
Brief Title: A Randomized Trial of the Rapamycin Target Eluting Stent for the Treatment of Symptomatic Cerebral Artery Atherosclerotic Disease（TARGET-DREAM）
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALIM-2024-01-CIP-00
Record Dates: First submitted 2025-03-27; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Intracranial Arteriosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental Group A（a self-expanding rapamycin target-eluting stent ） (Experimental): Approximately 83 subjects with symptomatic cerebral artery atherosclerotic stenosis will be enrolled in China and randomized to Experimental Group A（total 249 subjects in randomization group in China）
  Interventions: Device: Experimental Device A, a self-expanding rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China)
- Experimental Device B（a balloon-expandable rapamycin target-eluting stent） (Experimental): Approximately 83 subjects with symptomatic cerebral artery atherosclerotic stenosis will be enrolled in China and randomized to Experimental Group B（total 249 subjects in randomization group in China）
  Interventions: Device: Experimental Device B, a balloon-expandable rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China)
- Control group（Apollo® Intracranial Artery Stent System, a balloon-expandable bare-metal stent） (Active Comparator): Approximately 83 subjects with symptomatic cerebral artery atherosclerotic stenosis will be enrolled in China and randomized to control group（total 249 subjects in randomization group in China）
  Interventions: Device: Apollo® Intracranial Artery Stent System, a balloon-expandable bare-metal stent (MicroPort NeuroTech, Shanghai, China),
- Specification subgroup (Other): 20 subjects with lesions only suitable for the unique specifications of Experimental Device A or Experimental Device B will be enrolled in China. These subjects will not undergo randomization, and their data will be analyzed separately without hypothesis testing.
  Interventions: Device: Experimental Device A, a self-expanding rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China); Device: Experimental Device B, a balloon-expandable rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China)
- Overseas subgroup for Experimental Device B in Brazil (Other): A subgroup of Experimental Device B is established at a study center in Brazil. 10 subjects meeting the trial's inclusion and criteria will be enrolled. These subjects will not undergo randomization, and their data will be analyzed separately without hypothesis testing, only to support overseas registration
  Interventions: Device: Experimental Device B, a balloon-expandable rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China)

INTERVENTIONS:
Device: Experimental Device A, a self-expanding rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China) — Experimental Device A, a self-expanding rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China)
  Arms: Experimental Group A（a self-expanding rapamycin target-eluting stent ）; Specification subgroup
Device: Experimental Device B, a balloon-expandable rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China) — Experimental Device B, a balloon-expandable rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China)
  Arms: Experimental Device B（a balloon-expandable rapamycin target-eluting stent）; Overseas subgroup for Experimental Device B in Brazil; Specification subgroup
Device: Apollo® Intracranial Artery Stent System, a balloon-expandable bare-metal stent (MicroPort NeuroTech, Shanghai, China), — Apollo® Intracranial Artery Stent System, a balloon-expandable bare-metal stent (MicroPort NeuroTech, Shanghai, China)
  Arms: Control group（Apollo® Intracranial Artery Stent System, a balloon-expandable bare-metal stent）

SUMMARY:
The trial is a prospective, multicenter, open-label, superiority, randomized controlled clinical trial. The experimental groups include two types of drug-eluting stents:

* Experimental Device A, a self-expanding rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China)
* Experimental Device B, a balloon-expandable rapamycin target-eluting stent (MicroPort NeuroTech, Shanghai, China) The device used in the control group is the Apollo® Intracranial Artery Stent System, a balloon-expandable bare-metal stent (MicroPort NeuroTech, Shanghai, China), According to the inclusion and exclusion criteria specified in the protocol, approximately 249 subjects with symptomatic cerebral artery atherosclerotic stenosis will be enrolled in China and randomized to Experimental Group A, Experimental Group B, or the control group.

Considering the broader applicability of Experimental Device A and Experimental Device B compared to the control device, a specification subgroup is established. 20 subjects with lesions only suitable for the unique specifications of Experimental Device A or Experimental Device B will be enrolled in China. These subjects will not undergo randomization, and their data will be analyzed separately without hypothesis testing.

Moreover, a subgroup of Experimental Device B is established at a study center in Brazil. 10 subjects meeting the trial's inclusion and criteria will be enrolled. These subjects will not undergo randomization, and their data will be analyzed separately without hypothesis testing, only to support overseas registration.

Overall, the total sample size for the study is 279 subjects. Clinical assessment will be conducted for all subjects before the procedure, during the procedure, at discharge, at 1 month (±7 days) follow-up, at 6 months (±30 days) follow-up, and at 12 months (±60 days) follow-up. At 12 months (±60 days), patients will undergo follow-up with DSA imaging. Unscheduled follow-ups may be performed as needed to record relevant indicators and evaluate the safety and efficacy of the two drug-eluting stents in the treatment of symptomatic cerebral artery atherosclerotic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18-80 years old
* 2) Symptomatic cerebral artery atherosclerotic stenosis (defined as ischemic stroke or TIA due to qualifying lesion stenosis occurring in the past 6 months) with ineffective antiplatelet therapy or hypoperfusion in the territory of qualifying artery or with poor collateral circulation
* 3) Lesion located in a major cerebral artery, including the internal carotid artery, middle cerebral artery, vertebral artery, or basilar artery
* 4) 70%-99% stenosis of qualifying lesion according to WASID method diagnosed by DSA
* 5) Subject with at least one or more risk factors, including hypertension, diabetes mellitus, hyperlipidemia, hyperhomocysteinemia, coronary artery disease, obesity, smoking history, etc
* 6) Subject and/or their legal representatives have the necessary mental capacity to understand the study purpose, agree to participate in the study, and sign the informed consent form

Exclusion Criteria:

* 1) mRS score≥3
* 2) Last ischemic stroke onset within 2 weeks
* 3) Presence of 2 or more atherosclerotic stenotic lesions in the cerebral arteries requiring interventional or surgical treatment.
* 4) Only perforator infarctions in the territory of qualifying artery according to preoperative imaging
* 5) Hemorrhagic transformation in the territory of qualifying artery. Any parenchymal, subarachnoid, subdural, or extradural hemorrhage within 30 days prior to procedure, or untreated chronic subdural hematoma(≥5 mm) according to preoperative imaging
* 6) Restenosis of qualifying lesion due to previous stenting.
* 7) Qualifying lesion with severe calcification, extreme eccentricity, or extreme angulation which may affect stent deployment
* 8) Stenosis caused by non-atherosclerotic lesions, such as arterial dissection, moya-moya disease, or vasculitis
* 9) Concomitant severe stenosis (≥70% stenosis as measured by the WASID method) in the distal or proximal to qualifying lesion
* 10) Concomitant multiple stenoses where qualifying lesions cannot be identified
* 11) Thrombus in the qualifying artery or complete occlusion of the qualifying artery
* 12) Severe calcification or tortuosity of qualifying artery to prevent stent from successful positioning and dilatation
* 13) Stenting in qualifying artery within one year
* 14) Concomitant aneurysms requiring treatment
* 15) Concomitant intracranial malignant tumors, intracranial arteriovenous malformations, intracranial venous sinus thrombosis, or other conditions inappropriate to participate in the study
* 16) Resistant hypertension (systolic pressure ≥180 mmHg or diastolic pressure ≥110 mmHg) despite use of medication
* 17) Acute myocardial infarction within 4 weeks prior to enrollment, or suspected cardiogenic embolism
* 18) Subjects with severe systemic diseases that cannot tolerate surgery, such as severe hepatic or renal impairment
* 19) Severe cognitive impairment or mental diseases
* 20) Contraindications to anticoagulants or antiplatelet drugs, such as anticoagulant or antiplatelet drug allergy, active bleeding, or coagulation disorder
* 21) Subjects with allergy or suspected allergy to anesthetics, contrast agents, rapamycin, polylactic acid, nickel-titanium alloy, cobalt-chromium alloy, stainless steel, and other stent materials, medications, and intraoperative medications
* 22) Women who are pregnant or breastfeeding
* 23) Subjects who are participating or planning to participate in any drug or device clinical study at the time of enrollment
* 24) Life expectancy ≤ 1 year
* 25) Other conditions inapplicable to participate in the study according to investigators' judgment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
In-stent restenosis (ISR) rate at 12 months post-procedure | 12 months after surgery(±60days)
  ISR is defined as >50% stenosis within or adjacent (within 5 mm) to the stent as well as >20% absolute luminal loss according to the WASID method diagnosed by DSA

SECONDARY OUTCOMES:
Technical success rate of stent implantation | Day 0（within 1hour after procedure）
  defined as successful implantation into qualifying lesion as well as successful retraction of delivery system
Symptomatic ISR rate at 12 months post-procedure | 12 months after surgery(±60days)
  ISR (ISR is defined as >50% stenosis within or adjacent (within 5 mm) to the stent as well as >20% absolute luminal loss according to the WASID method diagnosed by DSA) occurs with ischemic stroke or TIA from target lesion restenosis.
  Stroke is defined as acute focal/systemic neurological dysfunction from brain/spinal cord/retinal vascular occlusion, stenosis, or injury - induced hemorrhage/infarction.
  TIA is defined as transient focal neurological dysfunction from brain/spinal cord/retinal ischemia, with symptoms lasting<24 hours and no acute infarction.
Revascularization rate from qualifying artery at 12 months post-procedure | During the days of follow-up(up to 12month ±60 days)
  During follow-up, revascularization procedures (including interventional thrombectomy, angioplasty, vascular bypass, etc.) due to ischemic stroke or TIA from target lesions.
  Stroke is defined as acute focal/systemic neurological dysfunction from brain/spinal cord/retinal vascular occlusion, stenosis, or injury - induced hemorrhage/infarction.
  TIA is defined as transient focal neurological dysfunction from brain/spinal cord/retinal ischemia, with symptoms lasting<24 hours and no acute infarction.
Modified Rankin Scale (mRS) score at 12 months post-procedure | 12 months after surgery(±60days)
Stroke or death related to qualifying lesion at 30 days, 6 months, and 12 months post-procedure | During the days of follow-up(up to 12month ±60 days)
  Stroke is defined as acute focal/systemic neurological dysfunction from brain/spinal cord/retinal vascular occlusion, stenosis, or injury - induced hemorrhage/infarction.
Any stroke or death at 30 days, 6 months, and 12 months post-procedure | During the days of follow-up(up to 12month ±60 days)
  Stroke is defined as acute focal/systemic neurological dysfunction from brain/spinal cord/retinal vascular occlusion, stenosis, or injury - induced hemorrhage/infarction.
Study device related serious adverse event rate during follow-up | During the days of follow-up(up to 12month ±60 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No